CLINICAL TRIAL: NCT01284257
Title: A Phase IV, Non-interventional, Multi-center, Open-label, Prospective, Observational Study of the Safety, Effectiveness, Tolerability and Compliance of Immunosuppressive Regimens Using Mycophenolic Acid to Treat de Novo Renal Transplant Patients in Routine Clinical Practice
Brief Title: Observational Registry Study of Renal Transplant Patients
Acronym: MORE registry
Status: Withdrawn | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CERL080AUS40
Record Dates: First submitted 2011-01-25; First posted 2011-01-26 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Kidney Transplant
Keywords: EC-MPS; MMF; kidney transplant; outcomes; mycophenolate sodium; mycophenolic acid (MPA)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Enteric coated mycophenolate sodium (EC-MPS) arm: Patients to whom EC-MPS is prescribed by their practitioner.
- MMF arm: Patients to whom MMF is prescribed by their practitioner.

SUMMARY:
The MORE Observational Study follows real-world renal transplant patients with the data resolution of a monitored, prospective clinical trial for 5 years. In addition to capturing detailed clinical data, the study describes recent important changes in surveillance testing and drug therapy and relates these changes to short and long-term outcomes. Also, the study measures patient compliance over time and details the rationale for modifications of MPA dosing in maintenance and regimen changes after episodes of AR. The MORE study will provide information on era changes in transplant practices and their impact on clinical outcome, new insights on optimizing regimens for discrete patient subsets and new perspectives on the optimal use of MPA therapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* The de novo recipient of a cadaveric or living donor kidney transplant, within two weeks of transplantation.
* Receiving mycophenolic acid (MPA) therapy of either myfortic® or CellCept®.
* Able to provide informed consent.
* Able to self-administer the ITAS compliance instrument (6 questions).

Exclusion Criteria:

* The recipient of multiple organ grafts or prior non-kidney graft.
* Enrolled or plans to enroll in an investigational clinical trial.
* Not likely to have up to 5 year follow-up data available for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll approximately 1,200 de novo (newly transplanted within 2 weeks) renal transplant patients from approximately 30-60 transplant centers across the United States. Patients should be consented prior to the first dose of MPA, +/- 14 days from the date of the transplant and be enrolled as soon as feasible after transplantation but not later than 2 weeks post-transplantation. Enrollment targets will be capped globally at 800 patients being treated with myfortic® and 400 patients being treated with CellCept®.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Dosage of EC-MPS or MMF over time | 60 months
  Dosage interruptions, discontinuations and switches between EC-MPS and MMF

SECONDARY OUTCOMES:
Incidence of Gastro-Intestinal (GI) Adverse Events (AEs) in relationship with prior GI history and GI co-medications | 60 months
The incidence of selected Adverse Events | 60 months
  e.g., viral infections, hematological events, glaucoma, malignancy, diabetes mellitus, cardiovascular events, bone-loss related events, GI events, hepatitis) and associated Serious Adverse Events (SAEs).
Combined outcome measure of biopsy-proven acute rejection (BPAR) episodes, graft loss and death | 60 months
Center Practices | 60 months
  The center practice will be described as observed. This includes the number of transplants performed per year per center, patient follow up frequency, performance of protocol biopsies, use of induction therapies and MPA monitoring.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - San Francisco investigational site, San Francisco, California
  - Denver Investigational site, Denver, Colorado
  - Springfield investigational site, Springfield, Massachusetts
  - Detroit investigational site, Detroit, Michigan
  - New York investigational site, New York, New York
  - PHILADELPHIA investigational site, Philadelphia, Pennsylvania
  - BURLINGTON investigational site, Burlington, Vermont
  - Seattle investigational site, Seattle, Washington